CLINICAL TRIAL: NCT03723005
Title: A Light Emitting Diode (LED) Mattress for Phototherapy of Jaundiced Newborns
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: NeoLight, LLC. (Unknown)
Responsible Party: Principal Investigator, David K Stevenson, PI, Stanford University
Other Study IDs: IRB-41341
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Neolight Phototherapy Mattress: Once a qualified patient is enrolled, he/she will be randomized to Neolight phototherapy or standard-of-care phototherapy, which is ordered by physician as part of routine. Duration of phototherapy exposure will be recorded as entered by RN in patient medical progress notes.
  Interventions: Device: Neolight Phototherapy Mattress
- Standard-of-Care Phototherapy: Once a qualified patient is enrolled, he/she will be randomized to Neolight phototherapy or standard-of-care phototherapy, which is ordered by physician as part of routine. Duration of phototherapy exposure will be recorded as entered by RN in patient medical progress notes.
  Interventions: Device: Standard-of-Care

INTERVENTIONS:
Device: Neolight Phototherapy Mattress — Once a qualified patient is enrolled, he/she will be randomized to Neolight phototherapy or standard-of-care phototherapy, which is ordered by physician as part of routine. Duration of phototherapy exposure will be recorded as entered by RN in patient medical progress notes.
  Groups: Neolight Phototherapy Mattress
Device: Standard-of-Care — Once a qualified patient is enrolled, he/she will be randomized to Neolight phototherapy or standard-of-care phototherapy, which is ordered by physician as part of routine. Duration of phototherapy exposure will be recorded as entered by RN in patient medical progress notes.
  Groups: Standard-of-Care Phototherapy

SUMMARY:
The new investigational and FDA-approved device is named "SkyLife" and is a mattress, which uses blue LEDs as the light source similar to those used in the currently-used overhead blue LED panel devices.

DETAILED DESCRIPTION:
The new investigational and FDA-approved device is named "SkyLife" and is a mattress, which uses blue LEDs as the light source similar to those used in the currently-used overhead blue LED panel devices. It is believed that this device will not only avoid many of the side effects when fluorescent tube lights are used, since it delivers safer, non-ultraviolet light; but may also be more effective than currently-used blankets or mattresses, which use blue halogen lamps or fluorescent tubes as light sources. The light is emitted under the baby. This study will discover if this device should be used in place of the currently-used devices.

ELIGIBILITY:
Inclusion Criteria:

* Male and female newborns greater of equal to 28 weeks GA
* Parental informed consent
* Enrollment at age greater than 6 hrs of age until neonatal discharge
* Phototherapy routine order

Exclusion Criteria:

* Infant requiring respiratory assistance (such as mechanical ventilation)
* Severe or life-threatening congenital anomalies
* Blood transfusion history

Ages: 28 Weeks to 8 Months | Sex: All
Age Groups: Child
Study Population: All infants (not gender or racial/ethnically based) equal or greater than 28 weeks GA and great than 6 hrs of age until hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Total Bilirubin (TB) Levels | up to 1 week
  Efficacy of each device (neoLight and conventional devices) will be assessed as a decrease in TB levels (in mg/dL/hr) for each infant in each study group
Duration of Phototherapy | up to 1 week
  Efficacy of each device (neoLight and conventional devices) will also be assessed as the duration (in hrs) of phototherapy for each infant in each study group.

SECONDARY OUTCOMES:
Irradiance Stability of the neoLight Device | 1 year
  The performance of the neoLight will be assessed as the stability of irradiance emitted by the neoLight device during the use of the device
Infant Temperature Change | up to 1 week
  Safety of the neoLight device will be assessed as no change in an infant's temperature during phototherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Wong, MD, Study Director — Investigator
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Sharable statistical data in regards to efficacy of device compared to Standard-of-care devices already used in a hospital setting.